CLINICAL TRIAL: NCT00146250
Title: Relationship of Oxygenation During Anaesthesia in the Presence of N2O or N2 to Mode of Ventilation
Brief Title: The Effect of N2O Administration on Arterial Oxygenation
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Austin Health (Other Government)
Collaborators: Monash University (Other); La Trobe University (Other); The Alfred (Other); University of Melbourne (Other)
Responsible Party: Principal Investigator, Dr Philip Peyton, Doctor, Austin Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H99/00835
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Anesthesia
MeSH Terms: interventions — Nitrous Oxide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Nitrous oxide (Experimental): Nitrous oxide 70% as balance gas in inspired mixture
  Interventions: Drug: Nitrous oxide
- Nitrogen (Experimental): Nitrogen instead of nitrous oxide 70% as balance gas in inspired mixture
  Interventions: Drug: Nitrous oxide

INTERVENTIONS:
Drug: Nitrous oxide — Substitution of Nitrous oxide for Nitrogen as balance gas in inspired gas mixture
  Other Names: N2O

SUMMARY:
Nitrous oxide is a standard part of most anaesthetic breathing mixtures. It has often been assumed that it reduces the amount of oxygen reaching the lower parts of the lung. However the results of previous studies and of some computer modelling suggests the opposite may be true, and that oxygen levels in the blood are actually higher with nitrous oxide. This study seeks to determine whether nitrous oxide increases or decreases blood oxygen levels in anaesthetized patients.

DETAILED DESCRIPTION:
The concentrating and second gas effects of nitrous oxide (N2O) uptake have been well described, and are produced by rapid uptake of N2O during the first several minutes of an inhalational anesthetic. This significantly increases alveolar and arterial O2 partial pressure. Theoretical modelling of alveolar gas exchange has predicted that these effects may not be transient but may be a persisting phenomenon. However, N2O is known to promote absorption atelectasis in poorly ventilated lung units.

This study, carried out pre-cardiopulmonary bypass in 20 patients undergoing coronary artery surgery, measures change in PaO2 after a minimum of 30 minutes of relaxant general anesthesia with a FIO2 of 30%. Patients are randomised to two groups. The intervention group has N2O introduced following baseline blood gas measurements, while the control group continued breathing an identical FIO2 in N2. The change in PaO2 in the two groups is the primary endpoint for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing elective coronary artery bypass surgery

Exclusion Criteria:

* Age under 18 years, emergency surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-03-01 (Actual); Primary Completion 2005-07-20 (Actual); Study Completion 2005-09-30 (Actual)

PRIMARY OUTCOMES:
PaO2 | Minimum of 30 minutes after induction of anaesthesia
  Measured change in PaO2 after a minimum of 30 minutes of general anaesthesia, following sternotomy, in the two groups.

SECONDARY OUTCOMES:
Change in pulmonary deadspace and shunt fractions | Minimum of 30 minutes after induction of anaesthesia
  Change in pulmonary deadspace and shunt fractions, as calculated by the Bohr and shunt equations.

CONTACTS AND LOCATIONS:
Overall Officials: Philip J Peyton, MD FANZCA, Principal Investigator — Dept of Anaesthesia, Austin Health